CLINICAL TRIAL: NCT00640315
Title: Proof of Concept Study to Investigate Safety, Tolerability, Pharmacokinetics and the Impact on Pulmonary and Systemic Hemodynamics, Gas Exchange and Lung Function Parameters of a Single-dose of BAY63-2521 IR-tablet in Patients With COPD Associated Pulmonary Hypertension in an Non-randomized, Non-blinded Design
Brief Title: Single Dose Study in Patients With Chronic Obstructive Pulmonary Disease (COPD) Associated Pulmonary Hypertension.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12915; 2007-003919-31 (EudraCT Number)
Record Dates: First submitted 2008-02-29; First posted 2008-03-21 (Estimated); Results first posted 2014-02-28 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-11

CONDITIONS: Hypertension, Pulmonary; Pulmonary Disease, Chronic Obstructive
Keywords: Chronic obstructive pulmonary disease; COPD; Pulmonary hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Disease, Chronic Obstructive | interventions — riociguat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Riociguat (Adempas, BAY63-2521) 1.0 mg (Experimental): Participants received two single oral doses of 1.0 mg riociguat on study day 1 and study day 3.
  Interventions: Drug: Riociguat (Adempas, BAY63-2521) 1.0 mg
- Riociguat (Adempas, BAY63-2521) 2.5 mg (Experimental): Participants received two single oral doses of 2.5 mg riociguat on study day 1 and study day 3.
  Interventions: Drug: Riociguat (Adempas, BAY63-2521) 2.5 mg

INTERVENTIONS:
Drug: Riociguat (Adempas, BAY63-2521) 1.0 mg — 1.0 mg BAY63-2521 will be given twice per subject, as single dose administration during the hemodynamic investigation (on study day 1) and during the lung function testing (on study day 3).
  Arms: Riociguat (Adempas, BAY63-2521) 1.0 mg
Drug: Riociguat (Adempas, BAY63-2521) 2.5 mg — 2.5 mg BAY63-2521 will be given twice per subject, as single dose administration during the hemodynamic investigation (on study day 1) and during the lung function testing (on study day 3).
  Arms: Riociguat (Adempas, BAY63-2521) 2.5 mg

SUMMARY:
This study is to demonstrate the safety, tolerability, pharmakokinetic and pharmacodynamic effect of a single oral dose of BAY63-2521 in patients with pulmonary hypertension due to chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
In addition to the pharmacodynamic and pharmacokinetic variables, the following laboratory variables were assessed:

* Hematology: Leucocytes, erythrocytes, hemoglobin, hematocrit, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), platelets, white blood cell (WBC), partial thromboplastin time (PTT), prothrombin time (Quick), international normalized ratio (INR) (prothrombin time expressed in relation to normal value) ;
* Clinical chemistry: aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (AP), gamma glutamyl transpeptidase (GGT), creatine phosphokinase (CK), lipase, cholinesterase (CHE), glucose, creatinine, urea, uric acid, bilirubin, total protein, serum albumin, sodium, potassium, calcium, chloride.

And due to the small number of subjects analyzed at several local labs, no summary statistics were provided.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pulmonary hypertension due to COPD, undergoing routine invasive measurement of hemodynamic parameters.
* Catheters for measurement of hemodynamic parameters (PAP [pulmonary artery pressure], PCWP [pulmonary capillary wedge pressure], CO [cardiac output], SBP [systolic blood pressure]) must be in place independent of the trial.

Exclusion Criteria:

* Acute exacerbation of COPD,
* Pre-existing lung disease other than COPD,
* Acute or severe chronic left heart failure,
* Severe coronary artery disease,
* Uncontrolled arterial hypertension;
* Severe left ventricular hypertrophy,
* Congenital or acquired valvular or myocardial disease,
* Systolic blood pressure < 100 mmHg,
* Heart rate < 55 bpm or >105 bpm,
* PaO2 (arterial partial oxygen pressure)/FiO2 (fraction of inspired oxygen) < 50 mmHg,
* PaCO2 (arterial partial pressure of carbon dioxide) > 55 mmHg,
* Severe hepatic insufficiency,
* Severe renal insufficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (7):
- Germany (7):
  - Heidelberg, Baden-Wurttemberg
  - Löwenstein, Baden-Wurttemberg
  - München, Bavaria
  - Bad Nauheim, Hesse
  - Giessen, Hesse
  - Greifswald, Mecklenburg-Vorpommern
  - Dresden, Saxony

REFERENCES:
- [Result] H.-A. Ghofrani, G. Staehler, E. Gruenig, M. Halank, V. Mitrovic, S. Unger, W. Mueck, R. Frey, J. Behr. The Effect Of The Soluble Guanylate Cyclase Stimulator Riociguat On Hemodynamics In Patients With Pulmonary Hypertension Due To Chronic Obstructive Pulmonary Disease. D96 CLINICAL TRIALS AND OUTCOMES IN PULMONARY HYPERTENSION.
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Started | 10 | 13
Participants Received Treatment | 10 | 13
Completed | 10 | 12
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg | Total
Number analyzed (Participants) | 10 | 13 | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.5 (8.9) [56 to 82] | 69.2 (5.7) [61 to 79] | 68.4 (7.1) [56 to 82]
Gender [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Swan-Ganz Hemodynamics - Maximal Change From Baseline at Day 1 of Mean Pulmonary Artery Pressure (PAPmean)
Description: PAPmean was reported during right heart catheterization
Time Frame: From baseline up to 4 hours after administration
Population: per-protocol population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 10 | 12
mmHg | -3.60 (3.41) | -4.83 (4.17)

2. Primary Outcome: Swan-Ganz Hemodynamics - Maximal Change From Baseline at Day 1 of Pulmonary Vascular Resistance (PVR)
Description: PVR was calculated according to the formula PVR = 80*(PAPmean - pulmonary capillary wedge pressure)/cardiac output
Time Frame: From baseline up to 4 hours after administration
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: (dyn*s*cm^-5)
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 10 | 11
(dyn*s*cm^-5) | -58.32 (50.46) | -123.8 (73.53)

3. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Zero to Infinity (AUC) of Riociguat and Metabolite M1 After Single Dose of Riociguat
Time Frame: Study day 1: 0, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 24, 36 hours post-dose; Study day 3: 0, 2, 6, 12, 24 hours post-dose
Population: per-protocol population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/L
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 10 | 12
µg*h/L
  Riociguat - Study day 1 (00d01h) | 481.9 (65.3) | 1319 (56.8)
  Riociguat - Study day 3 (02d01h) | 605.5 (79.1) | 999.5 (61.6)
  Metabolite M1 - Study day 1 (00d01h) | NA (NA) — Insufficient number of participants with data. | 1019 (26.0)
  Metabolite M1 - Study day 3 (02d01h) | NA (NA) — Insufficient number of participants with data. | NA (NA) — Insufficient number of participants with data.

4. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Zero to Infinity Divided by Dose (AUC/D) of Riociguat and Metabolite M1 After Single Dose of Riociguat
Time Frame: Study day 1: 0, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 24, 36 hours post-dose; Study day 3: 0, 2, 6, 12, 24 hours post-dose
Population: per-protocol population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 10^3*h/L
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 10 | 12
10^3*h/L
  Riociguat - Study day 1 (00d01h) | 481.9 (65.3) | 527.4 (56.8)
  Riociguat - Study day 3 (02d01h) | 605.5 (79.1) | 399.8 (61.6)
  Metabolite M1 - Study day 1 (00d01h) | NA (NA) — Insufficient number of participants with data. | 421.6 (26.0)
  Metabolite M1 - Study day 3 (02d01h) | NA (NA) — Insufficient number of participants with data. | NA (NA) — Insufficient number of participants with data.

5. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Zero to Infinity Divided by Dose Per kg Body Weight (AUCnorm) of Riociguat and Metabolite M1 After Single Dose of Riociguat
Time Frame: Study day 1: 0, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 24, 36 hours post-dose; Study day 3: 0, 2, 6, 12, 24 hours post-dose
Population: per-protocol population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: kg*h/L
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 10 | 12
kg*h/L
  Riociguat - Study day 1 (00d01h) | 35.53 (62.6) | 38.85 (56.7)
  Riociguat - Study day 3 (02d01h) | 44.86 (68.0) | 29.93 (65.7)
  Metabolite M1 - Study day 1 (00d01h) | NA (NA) — Insufficient number of participants with data. | 31.03 (27.1)
  Metabolite M1 - Study day 3 (02d01h) | NA (NA) — Insufficient number of participants with data. | NA (NA) — Insufficient number of participants with data.

6. Primary Outcome: Maximum Drug Concentration in Plasma (Cmax) of Riociguat and Metabolite M1 After Single Dose of Riociguat
Time Frame: Study day 1: 0, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 24, 36 hours post-dose; Study day 3: 0, 2, 6, 12, 24 hours post-dose
Population: per-protocol population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/L
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 10 | 12
µg/L
  Riociguat - Study day 1 (00d01h) | 42.96 (32.3) | 116.0 (36.0)
  Riociguat - Study day 3 (02d01h) | 35.30 (46.0) | 80.44 (27.3)
  Metabolite M1 - Study day 1 (00d01h) | 10.44 (56.5) | 27.27 (34.9)
  Metabolite M1 - Study day 3 (02d01h) | 9.869 (37.2) | 26.49 (26.5)

7. Primary Outcome: Maximum Drug Concentration in Plasma Divided by Dose (Cmax/D) of Riociguat and Metabolite M1 After Single Dose of Riociguat
Time Frame: Study day 1: 0, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 24, 36 hours post-dose; Study day 3: 0, 2, 6, 12, 24 hours post-dose
Population: per-protocol population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 10^3/L
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 10 | 12
10^3/L
  Riociguat - Study day 1 (00d01h) | 42.96 (32.3) | 46.42 (36.0)
  Riociguat - Study day 3 (02d01h) | 35.30 (46.0) | 32.18 (27.3)
  Metabolite M1 - Study day 1 (00d01h) | 10.80 (56.5) | 11.28 (34.9)
  Metabolite M1 - Study day 3 (02d01h) | 10.21 (37.2) | 10.96 (26.5)

8. Primary Outcome: Maximum Drug Concentration in Plasma Divided by Dose Per kg Body Weight (Cmax,Norm) of Riociguat and Metabolite M1 After Single Dose of Riociguat
Time Frame: Study day 1: 0, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 24, 36 hours post-dose; Study day 3: 0, 2, 6, 12, 24 hours post-dose
Population: per-protocol population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: kg/L
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 10 | 12
kg/L
  Riociguat - Study day 1 (00d01h) | 3.185 (27.0) | 3.419 (30.9)
  Riociguat - Study day 3 (02d01h) | 2.617 (39.1) | 2.370 (31.4)
  Metabolite M1 - Study day 1 (00d01h) | 0.800 (46.8) | 0.831 (31.7)
  Metabolite M1 - Study day 3 (02d01h) | 0.757 (26.8) | 0.807 (27.5)

9. Secondary Outcome: Swan-Ganz Hemodynamics - Maximal Change From Baseline at Day 1 of Mean Right Atrial Pressure (RAPmean)
Description: RAPmean was reported during right heart catheterization
Time Frame: From baseline up to 4 hours after administration
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 9 | 11
mmHg | -2.00 (1.41) | -0.64 (1.69)

10. Secondary Outcome: Swan-Ganz Hemodynamics - Maximal Change From Baseline at Day 1 of Systolic Pulmonary Artery Pressure (PAPsyst)
Description: PAPsyst was acquired during right heart catheterization
Time Frame: From baseline up to 4 hours after administration
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 10 | 12
mmHg | -6.90 (4.86) | -9.42 (6.73)

11. Secondary Outcome: Swan-Ganz Hemodynamics - Maximal Change From Baseline at Day 1 of Diastolic Pulmonary Artery Pressure (PAPdiast)
Description: PAPdiast was acquired during right heart catheterization
Time Frame: From baseline up to 4 hours after administration
Population: per-protocol population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 10 | 12
mmHg | -3.80 (4.73) | -3.25 (2.83)

12. Secondary Outcome: Swan-Ganz Hemodynamics - Maximal Change From Baseline at Day 1 of Pulmonary Capillary Wedge Pressure (PCWP)
Description: PCWP was acquired during right heart catheterization
Time Frame: From baseline up to 4 hours after administration
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 10 | 12
mmHg | -3.60 (3.57) | -1.17 (3.38)

13. Secondary Outcome: Swan-Ganz Hemodynamics - Maximal Change From Baseline at Day 1 of Heart Rate (HR)
Description: HR was acquired during right heart catheterization
Time Frame: From baseline up to 4 hours after administration
Population: per-protocol population
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 10 | 12
beats per minute | 9.40 (7.31) | 13.92 (8.68)

14. Secondary Outcome: Swan-Ganz Hemodynamics - Maximal Change From Baseline at Day 1 of Systolic Blood Pressure (SBP)
Description: Systolic arterial blood pressure was acquired during right heart catheterization.
Time Frame: From baseline up to 4 hours after administration
Population: per-protocol population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 10 | 12
mmHg | -26.30 (16.63) | -22.17 (15.24)

15. Secondary Outcome: Swan-Ganz Hemodynamics - Maximal Change From Baseline at Day 1 of Diastolic Blood Pressure (DBP)
Description: Diastolic arterial blood pressure was acquired during right heart catheterization.
Time Frame: From baseline up to 4 hours after administration
Population: per-protocol population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 10 | 12
mmHg | -13.50 (6.84) | -11.25 (9.50)

16. Secondary Outcome: Swan-Ganz Hemodynamics - Maximal Change From Baseline at Day 1 of Mean Arterial Pressure (MAP)
Description: MAP was acquired during right heart catheterization
Time Frame: From baseline up to 4 hours after administration
Population: per-protocol population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 10 | 12
mmHg | -17.10 (7.71) | -13.92 (8.03)

17. Secondary Outcome: Swan-Ganz Hemodynamics - Maximal Change From Baseline at Day 1 of Cardiac Output (CO)
Description: CO was measured in triplicate by the thermodilution technique
Time Frame: From baseline up to 4 hours after administration
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 10 | 11
L/min | 0.66 (0.48) | 1.61 (1.49)

18. Secondary Outcome: Swan-Ganz Hemodynamics - Maximal Change From Baseline at Day 1 of Pulmonary Vascular Resistance Index (PVRI)
Description: PVRI was calculated as PVRI = (80*(PAPmean - PCWP)/CO)*body surface area
Time Frame: From baseline up to 4 hours after administration
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: dyn*s*cm^-5*m^2
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 10 | 11
dyn*s*cm^-5*m^2 | -108.6 (93.46) | -222.1 (130.69)

19. Secondary Outcome: Swan-Ganz Hemodynamics - Maximal Change From Baseline at Day 1 of Systemic Vascular Resistance (SVR)
Description: SVR was calculated as SVR = 80*(MAP-RAPmean)/CO
Time Frame: From baseline up to 4 hours after administration
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: dyn*s*cm^-5
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 9 | 10
dyn*s*cm^-5 | -440.0 (205.78) | -467.7 (154.94)

20. Secondary Outcome: Swan-Ganz Hemodynamics - Maximal Change From Baseline at Day 1 of Systemic Vascular Resistance Index (SVRI)
Description: SVRI was calculated as SVRI = (80*(MAP - RAPmean)/CO)*body surface area
Time Frame: From baseline up to 4 hours after administration
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: dyn*s*cm^-5*m^2
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 9 | 10
dyn*s*cm^-5*m^2 | -836.4 (385.92) | -837.9 (276.17)

21. Secondary Outcome: Swan-Ganz Hemodynamics - Maximal Change From Baseline at Day 1 of Cardiac Index
Description: Cardiac index was calculated as cardiac index = CO / body surface area.
Time Frame: From baseline up to 4 hours after administration
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 10 | 11
L/min/m^2 | 0.35 (0.26) | 0.89 (0.83)

22. Secondary Outcome: Blood Gas Analysis - Percentage Change From Baseline at 2 Hours Post Dose of Arterial Partial Oxygen Pressure (PaO2)
Description: Arterial blood gas analysis was performed by insertion of an indwelling arterial cannula. Percent change was calculated as "100%*(value post dose - value at baseline)/ value at baseline".
Time Frame: Baseline and 2 hours post dose
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 10 | 9
Percentage | -12.64 (24.79) | -12.99 (14.00)

23. Secondary Outcome: Blood Gas Analysis - Percentage Change From Baseline at 2 Hours Post Dose of Arterial Partial Pressure of Carbon Dioxide (PaCO2)
Description: as for outcome 22
Time Frame: Baseline and 2 hours post dose
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 10 | 9
Percentage | 4.43 (20.93) | 4.04 (13.27)

24. Secondary Outcome: Blood Gas Analysis - Percentage Change From Baseline at 2 Hours Post Dose of Venous Oxygen Pressure (PvO2)
Description: Percent change was calculated as "100%*(value post dose - value at baseline)/ value at baseline".
Time Frame: Baseline and 2 hours post dose
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 10 | 6
Percentage | 0.87 (8.57) | 12.07 (10.53)

25. Secondary Outcome: Blood Gas Analysis - Percentage Change From Baseline at 2 Hours Post Dose of Arterial Oxygen Saturation (SaO2)
Description: as for outcome 22
Time Frame: Baseline and 2 hours post dose
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 10 | 9
Percentage | -2.23 (3.89) | -2.89 (3.84)

26. Secondary Outcome: Blood Gas Analysis - Percentage Change From Baseline at 2 Hours Post Dose of Venous Oxygen Saturation (SvO2)
Description: Percent change was calculated as "100%*(value post dose - value at baseline)/ value at baseline".
Time Frame: Baseline and 2 hours post dose
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 10 | 7
Percentage | 0.27 (6.58) | 6.76 (6.10)

27. Secondary Outcome: Lung Function - Percentage Change From Baseline at 2 Hours Post Dose of Forced Expiratory Volume in 1 Second (FEV1)
Time Frame: Baseline and 2 hours post dose
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 9 | 11
Percentage | 2.90 (3.32) | 3.81 (11.55)

28. Secondary Outcome: Lung Function - Percentage Change From Baseline at 2 Hours Post Dose of Percent of Predicted FEV1
Time Frame: Baseline and 2 hours post dose
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 9 | 11
Percentage | 3.00 (3.38) | 4.35 (11.88)

29. Secondary Outcome: Lung Function - Percentage Change From Baseline at 2 Hours Post Dose of Forced Vital Capacity (FVC)
Time Frame: Baseline and 2 hours post dose
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 9 | 11
Percentage | 5.16 (16.08) | 8.62 (23.73)

30. Secondary Outcome: Lung Function - Percentage Change From Baseline at 2 Hours Post Dose of Percent of Predicted FVC
Time Frame: Baseline and 2 hours post dose
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 8 | 11
Percentage | 0.41 (8.01) | 8.65 (23.77)

31. Secondary Outcome: Lung Function - Percentage Change From Baseline at 2 Hours Post Dose of FEV1/FVC
Time Frame: Baseline and 2 hours post dose
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 9 | 11
Percentage | -0.69 (11.26) | -1.29 (17.98)

32. Secondary Outcome: Lung Function - Percentage Change From Baseline at 2 Hours Post Dose of Total Lung Capacity (TLC)
Time Frame: Baseline and 2 hours post dose
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 9 | 10
Percentage | 1.86 (10.53) | 2.14 (10.85)

33. Secondary Outcome: Lung Function - Percentage Change From Baseline at 2 Hours Post Dose of Percent of Predicted TLC
Description: The percent of predicted TLC was provided by investigator at site.
Time Frame: Baseline and 2 hours post dose
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 9 | 10
Percentage | 1.91 (10.63) | 2.08 (10.92)

34. Secondary Outcome: Lung Function - Percentage Change From Baseline at 2 Hours Post Dose of Residual Volume (RV)
Time Frame: Baseline and 2 hours post dose
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 9 | 10
Percentage | 0.80 (9.15) | 3.16 (22.39)

35. Secondary Outcome: Lung Function - Percentage Change From Baseline at 2 Hours Post Dose of Percent of Predicted RV
Time Frame: Baseline and 2 hours post dose
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 9 | 10
Percentage | 0.83 (9.09) | 3.21 (22.46)

36. Secondary Outcome: Lung Function - Percentage Change From Baseline at 2 Hours Post Dose of Maximal Expiratory Flow at 75% of Expiratory Vital Capacity (MEF75)
Time Frame: Baseline and 2 hours post dose
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 7 | 11
Percentage | -0.92 (22.28) | -1.09 (17.38)

37. Secondary Outcome: Lung Function - Percentage Change From Baseline at 2 Hours Post Dose of Maximal Expiratory Flow at 50% of Expiratory Vital Capacity (MEF50)
Time Frame: Baseline and 2 hours post dose
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 9 | 10
Percentage | 0.17 (18.29) | 5.59 (15.03)

38. Secondary Outcome: Lung Function - Percentage Change From Baseline at 2 Hours Post Dose of Maximal Expiratory Flow at 25% of Expiratory Vital Capacity (MEF25)
Time Frame: Baseline and 2 hours post dose
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 8 | 8
Percentage | 8.56 (29.57) | -0.61 (40.44)

39. Secondary Outcome: Lung Function - Percentage Change From Baseline at 2 Hours Post Dose of Total Airway Resistance (Raw)
Time Frame: Baseline and 2 hours post dose
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 9 | 9
Percentage | -5.78 (24.03) | -5.89 (34.27)

40. Secondary Outcome: Lung Function - Percentage Change From Baseline at 2 Hours Post Dose of Vital Capacity (VC)
Time Frame: Baseline and 2 hours post dose
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 9 | 11
Percentage | 7.55 (22.35) | 10.09 (20.50)

41. Secondary Outcome: Lung Function - Percentage Change From Baseline at 2 Hours Post Dose of Percent of Predicted VC
Time Frame: Baseline and 2 hours post dose
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 9 | 11
Percentage | 7.60 (22.89) | 10.00 (20.45)

42. Secondary Outcome: Lung Function - Percentage Change From Baseline at 2 Hours Post Dose of Diffusing Capacity of the Lung for Carbon Monoxide (DLCO)
Time Frame: Baseline and 2 hours post dose
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 7 | 5
Percentage | 15.67 (26.65) | 18.66 (17.39)

43. Secondary Outcome: Lung Function - Percentage Change From Baseline at 2 Hours Post Dose of Total Lung Capacity at the Time When the DLCO is Measured (Alveolar Volume, VA)
Time Frame: Baseline and 2 hours post dose
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 7 | 4
Percentage | -2.35 (6.90) | 1.72 (12.79)

44. Secondary Outcome: Lung Function - Percentage Change From Baseline at 2 Hours Post Dose of Specific Diffusing Capacity
Time Frame: Baseline and 2 hours post dose
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 8 | 4
Percentage | 20.77 (27.36) | 18.61 (16.49)

45. Secondary Outcome: Multiple Inert Gas Elimination Technique (MIGET) Analysis - Change From Baseline at 1 Hour Post Dose of Total Ventilation (V)
Time Frame: Baseline and 1 hour post dose
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 5 | 2
L/min | -0.90 (1.00) | -0.10 (0.20)

46. Secondary Outcome: Multiple Inert Gas Elimination Technique (MIGET) Analysis - Change From Baseline at 1 Hour Post Dose of Total Perfusion (Q)
Time Frame: Baseline and 1 hour post dose
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 5 | 2
L/min | 0.30 (0.50) | -0.40 (0.50)

47. Secondary Outcome: Multiple Inert Gas Elimination Technique (MIGET) Analysis - Change From Baseline at 1 Hour Post Dose of Dead Space Ventilation
Time Frame: Baseline and 1 hour post dose
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: Percentage of total ventilation
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 5 | 1
Percentage of total ventilation | 3.20 (8.50) | -42.50 (NA) — n=1

48. Secondary Outcome: Multiple Inert Gas Elimination Technique (MIGET) Analysis - Change From Baseline at 1 Hour Post Dose of Low V/Q Perfusion
Time Frame: Baseline and 1 hour post dose
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 4 | 1
Percentage | 3.00 (13.40) | -0.30 (NA) — n=1

49. Secondary Outcome: Multiple Inert Gas Elimination Technique (MIGET) Analysis - Change From Baseline at 1 Hour Post Dose of Normal V/Q Perfusion
Time Frame: Baseline and 1 hour post dose
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 5 | 1
Percentage | -9.80 (21.00) | 4.10 (NA) — n=1

50. Secondary Outcome: Multiple Inert Gas Elimination Technique (MIGET) Analysis - Change From Baseline at 1 Hours Post Dose of Ventilation-perfusion Distribution Presented as Standard Deviation (SD) of Perfusion
Time Frame: Baseline and 1 hour post dose
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: L/MIN
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 5 | 1
L/MIN | 0.00 (0.10) | -0.10 (NA) — n=1

51. Secondary Outcome: Multiple Inert Gas Elimination Technique (MIGET) Analysis - Change From Baseline at 1 Hour Post Dose of Ventilation-perfusion Distribution Presented as Standard Deviation (SD) of Ventilation
Time Frame: Baseline and 1 hour post dose
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: L/MIN
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 5 | 1
L/MIN | -0.10 (0.40) | -0.50 (NA) — n=1

52. Secondary Outcome: Multiple Inert Gas Elimination Technique (MIGET) Analysis - Change From Baseline at 1 Hour Post Dose of Intrapulmonary Shunt Flow
Time Frame: Baseline and 1 hour post dose
Population: per-protocol population (subjects with data available for this outcome measure)
Measure: Mean (Standard Deviation); unit: Percentage of total perfusion
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 5 | 1
Percentage of total perfusion | -1.10 (1.70) | -0.30 (NA) — n=1

53. Secondary Outcome: Time to Reach Maximum Drug Concentration in Plasma (Tmax) of Riociguat and Metabolite M1 After Single Dose of Riociguat
Time Frame: Study day 1: 0, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 24, 36 hours post-dose; Study day 3: 0, 2, 6, 12, 24 hours post-dose
Population: per-protocol population
Measure: Median (Full Range); unit: hour
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 10 | 12
hour
  Riociguat - Study day 1 (00d01h) | 1.75 [0.917 to 4] | 1.742 [1 to 7.75]
  Riociguat - Study day 3 (02d01h) | 2.033 [2 to 5.917] | 2.042 [1.867 to 24.83]
  Metabolite M1 - Study day 1 (00d01h) | 11.97 [4 to 36.25] | 10.04 [3 to 24.33]
  Metabolite M1 - Study day 3 (02d01h) | 9.017 [2.15 to 24.42] | 12.04 [2 to 24.03]

54. Secondary Outcome: Half-life Associated With the Terminal Slope (t1/2) of Riociguat and Metabolite M1 After Single Dose of Riociguat
Time Frame: Study day 1: 0, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 24, 36 hours post-dose; Study day 3: 0, 2, 6, 12, 24 hours post-dose
Population: per-protocol population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 10 | 12
hour
  Riociguat - Study day 1 (00d01h) | 8.422 (58.6) | 9.541 (50.7)
  Riociguat - Study day 3 (02d01h) | 12.18 (47.5) | 8.835 (50.8)
  Metabolite M1 - Study day 1 (00d01h) | NA (NA) — Insufficient number of participants with data. | 20.57 (46.4)
  Metabolite M1 - Study day 3 (02d01h) | NA (NA) — Insufficient number of participants with data. | NA (NA) — Insufficient number of participants with data.

55. Secondary Outcome: Mean Residence Time (MRT) of Riociguat and Metabolite M1 After Single Dose of Riociguat
Time Frame: Study day 1: 0, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 24, 36 hours post-dose; Study day 3: 0, 2, 6, 12, 24 hours post-dose
Population: per-protocol population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 10 | 12
hour
  Riociguat - Study day 1 (00d01h) | 12.92 (50.2) | 13.97 (46.5)
  Riociguat - Study day 3 (02d01h) | 18.88 (39.5) | 13.37 (46.5)
  Metabolite M1 - Study day 1 (00d01h) | NA (NA) — Insufficient number of participants with data. | 34.77 (41.1)
  Metabolite M1 - Study day 3 (02d01h) | NA (NA) — Insufficient number of participants with data. | NA (NA) — Insufficient number of participants with data.

56. Secondary Outcome: Area Under the Plasma Concentration Verse Time Curve From Zero to the Last Data Point (AUC0-tn) of Riociguat and Metabolite M1 After Single Dose of Riociguat
Time Frame: Study day 1: 0, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 24, 36 hours post-dose; Study day 3: 0, 2, 6, 12, 24 hours post-dose
Population: per-protocol population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/L
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 10 | 12
µg*h/L
  Riociguat - Study day 1 (00d01h) | 426.3 (66.1) | 1196 (55.8)
  Riociguat - Study day 3 (02d01h) | 294.7 (81.6) | 750.3 (41.3)
  Metabolite M1 - Study day 1 (00d01h) | 200.1 (76.6) | 727.4 (20.1)
  Metabolite M1 - Study day 3 (02d01h) | 139.4 (98.8) | 490.6 (29.1)

57. Other Pre Specified Outcome: Mean PR Duration (PRmean) - Change From Baseline to Day 3
Description: PR duration was evaluated as part of the 12-lead electrocardiogram. ECGs were recorded after the participant had been at rest for 15 minutes in a supine position.
Time Frame: Baseline and day 3
Population: All subjects who received at least one dose of the trial medication were included in the safety evaluation.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 8 | 6
msec | 0.64 (21.60) | 11.20 (27.57)

58. Other Pre Specified Outcome: Mean QRS Duration (QRSmean) - Change From Baseline to Day 3
Description: QRS duration was evaluated as part of the 12-lead electrocardiogram. ECGs were recorded after the participant had been at rest for 15 minutes in a supine position.
Time Frame: Baseline and day 3
Population: All subjects who received at least one dose of the trial medication were included in the safety evaluation.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 8 | 8
msec | -2.56 (5.79) | 0.68 (12.99)

59. Other Pre Specified Outcome: Mean QT Duration (QTmean) - Change From Baseline to Day 3
Description: QT duration was evaluated as part of the 12-lead electrocardiogram. ECGs were recorded after the participant had been at rest for 15 minutes in a supine position.
Time Frame: Baseline and day 3
Population: All subjects who received at least one dose of the trial medication were included in the safety evaluation.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 6 | 4
msec | -2.00 (22.03) | -36.88 (15.48)

60. Other Pre Specified Outcome: Mean QTcB Duration (Bazett's Correction Formula, QTcB) - Change From Baseline to Day 3
Description: Bazett-corrected QTcB duration was evaluated as part of the 12-lead electrocardiogram. ECGs were recorded after the participant had been at rest for 15 minutes in a supine position.
Time Frame: Baseline and day 3
Population: All subjects who received at least one dose of the trial medication were included in the safety evaluation.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 6 | 4
msec | -1.45 (23.08) | 0.95 (13.49)

61. Other Pre Specified Outcome: Mean QTcF Duration (Fridericia's Correction Formula, QTcF) - Change From Baseline to Day 3
Description: Fridericia-corrected QTcF duration was evaluated as part of the 12-lead electrocardiogram. ECGs were recorded after the participant had been at rest for 15 minutes in a supine position.
Time Frame: Baseline and day 3
Population: All subjects who received at least one dose of the trial medication were included in the safety evaluation.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Number analyzed (Participants) | 6 | 4
msec | -1.58 (20.15) | -12.73 (10.50)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected after signing the informed consent until 30 days after end of study treatment.
Arm/Group | Riociguat (Adempas, BAY63-2521) 1.0 mg | Riociguat (Adempas, BAY63-2521) 2.5 mg
Serious Adverse Events (participants affected / at risk) | 0/10 | 2/13
Other Adverse Events (participants affected / at risk) | 4/10 | 6/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Riociguat (Adempas, BAY63-2521) 1.0 mg (N=10) | Riociguat (Adempas, BAY63-2521) 2.5 mg (N=13)
Pneumonia (Infections and infestations) | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Riociguat (Adempas, BAY63-2521) 1.0 mg (N=10) | Riociguat (Adempas, BAY63-2521) 2.5 mg (N=13)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
C-reactive protein increased (Investigations) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator may prepare the data derived from the Trial for publication. Such data will be submitted to the Sponsor for review at least 60 days prior to submission for publication. The Sponsor should respond within 50 days after receipt of the manuscript. The Investigator agrees that all reasonable comments made by the Sponsor in relation to a proposed publication will be incorporated. Confidential data provided by the Sponsor may not be published without written approval of the Sponsor.